CLINICAL TRIAL: NCT00579501
Title: A Multicenter Phase II Clinical Trial of Neoadjuvant Trabectedin (Yondelis) in Patients With Localized Myxoid / Round Cell Liposarcoma
Brief Title: Safety and Efficacy Study of Trabectedin for the Treatment of Localized Myxoid / Round Cell Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014767; ET-B-028-06 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Liposarcoma,Myxoid
Keywords: Myxoid; Liposarcoma; Trabectedin; Dexamethasone
MeSH Terms: conditions — Liposarcoma, Myxoid; Liposarcoma | interventions — Trabectedin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trabectedin (Experimental): Trabectedin at a dose of 1.5 milligram per meter square (mg/m^2) will be given as an intravenous (iv) infusion (a fluid or a medicine delivered into a vein by way of a needle) over 24-hour every 3 weeks for a minimum of 3 and a maximum of 6 cycles prior to definitive surgery. Dexamethasone 20 mg iv will also be administered within 30 minutes before start of each trabectedin infusion.
  Interventions: Drug: Trabectedin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Trabectedin — Trabectedin 1.5 mg/m^2 over a 24-hour iv infusion every 3 weeks for a minimum of 3 and a maximum of 6 cycles of trabectedin.
Drug: Dexamethasone — Dexamethasone 20 mg iv will be administered within 30 minutes before start of each trabectedin iv infusion

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of trabectedin for the treatment of localized (non-metastatic) myxoid / round cell liposarcoma (malignant tumor derived from primitive or embryonal lipoblastic cells).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), multicenter (when more than one hospital or medical school team work on a medical research study) study of trabectedin for the treatment of localized myxoid / round cell liposarcoma (MRCL). Trabectedin will be given at 1.5 milligram per meter square (mg/m^2) over a 24-hour intravenous (iv) infusion every 3 weeks for a minimum of 3 and a maximum of 6 cycles along with dexamethasone 20 mg iv which will be given within 30 minutes before start of each trabectedin iv infusion. Participants whose myxoid/round cell liposarcoma (MRCL) do not progress at the end of the neoadjuvant treatment will be followed every 6 weeks for disease progression or until 6 months post definitive surgery, in the absence of unacceptable toxicity and/or disease progression. Efficacy will be assessed by determining the pathologic Complete Response (pCR) rate assessed in the tumor surgical specimen by a central pathology review. Participants' safety will be monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of myxoid / round cell liposarcoma (MRCL) and availability of pathology specimens for central review and pharmacogenomic studies
* Clinical evidence of locally advanced (Stage III), non-metastatic tumor, including locally recurring disease after initial surgery
* Measurable disease (by Response Evaluation Criteria In Solid Tumors [RECIST])
* No prior chemotherapy or radiation (except for adjuvant post-operative radiotherapy)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2

Exclusion Criteria:

* Known hypersensitivity to any of the components of the trabectedin intravenous (iv) formulation or dexamethasone
* Pregnant or lactating women and women of reproductive potential who are not using effective contraceptive methods
* History of another neoplastic disease (except basal cell carcinoma or cervical carcinoma in situ adequately treated) unless in remission for 5 years or longer
* Known distant metastases
* Other serious illnesses such as congestive heart failure or angina pectoris, myocardial infarction within 1 year before enrollment, uncontrolled arterial hypertension or arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (8):
- United States (4):
  - Coeur d'Alene, Idaho
  - Park Ridge, Illinois
  - Iowa City, Iowa
  - Boston, Massachusetts
- France (3):
  - Bourdeaux
  - Lyon
  - Villejuif
- Mannheim, Germany

REFERENCES:
- [Derived] Gronchi A, Bui BN, Bonvalot S, Pilotti S, Ferrari S, Hohenberger P, Hohl RJ, Demetri GD, Le Cesne A, Lardelli P, Perez I, Nieto A, Tercero JC, Alfaro V, Tamborini E, Blay JY. Phase II clinical trial of neoadjuvant trabectedin in patients with advanced localized myxoid liposarcoma. Ann Oncol. 2012 Mar;23(3):771-776. doi: 10.1093/annonc/mdr265. Epub 2011 Jun 3. PMID 21642514

RESULTS

PARTICIPANT FLOW:
Groups:
- Trabectedin: Trabectedin at a dose of 1.5 milligram per meter square (mg/m^2) was given as an intravenous (iv) infusion (a fluid or a medicine delivered into a vein by way of a needle) over 24-hour every 3 weeks for a minimum of 3 and a maximum of 6 cycles prior to definitive surgery. Dexamethasone 20 mg iv was also administered within 30 minutes before start of each trabectedin infusion.
Period: Overall Study
Arm/Group | Trabectedin
Started | 29
Completed | 0
Not Completed | 29
Not completed — Death | 1
Not completed — End of neoadjuvant therapy | 25
Not completed — toxicity | 1
Not completed — Secondary lesion | 1
Not completed — Radiation therapy before surgery | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trabectedin
Number analyzed (Participants) | 29
Age, Customized [Number; unit: participants]
  18-49 years | 15
  50-69 years | 10
  greater than or equal to 70 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: Complete pathological response is complete disappearance of the tumor tissue up to the molecular level.
Time Frame: Every 6 weeks until disease progression (up to Week 33) or 6 months post surgery.
Population: Participants who received at least one cycle of trabectedin and have adequate pre and post trabectedin pathologic specimens available. Six participants were non evaluable for pCR assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Trabectedin
Number analyzed (Participants) | 23
percentage of participants | 13

2. Secondary Outcome: Percentage of Participants With Objective Tumor Response Based on Response Evaluation Criteria In Solid Tumors (RECIST)
Description: The objective tumor response is defined as the percentage of participants achieving partial response (PR) on tumor response assessed by RECIST. The PR is at least 30 percent decrease in sum of the longest diameter of target lesions or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Every 6 weeks until disease progression (up to Week 33) or 6 months post surgery.
Population: Participants who received at least one cycle of trabectedin and have at least one post baseline disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Trabectedin
Number analyzed (Participants) | 29
percentage of participants | 24.1

ADVERSE EVENTS:
Arm/Group | Trabectedin
Serious Adverse Events (participants affected / at risk) | 6/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=29)
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin (N=29)
Anaemia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 14
Bradycardia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Ventricular extrasystoles (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 3
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 22
Reflux gastritis (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 19
Infusion site pain (General disorders) | 2
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pyrexia (General disorders) | 8
Hepatotoxicity (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Injection site infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 2
Thrombophlebitis superficial (Vascular disorders) | 1
Headache (Nervous system disorders) | 5
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before submitting the paper or abstract or disclose information to public concerning trabectedin (YONDELIS®), PharmaMar must be provided of 15 days in case of abstract and 30 days in case of full paper, to review and approve the publication to assure that confidential and proprietary data are protected. Primary authorship for publication is hold by the coordinating investigator of this project. Following authors will be named according to the number of patients treated under this protocol.